CLINICAL TRIAL: NCT00815347
Title: The Effect of the ET-1 Receptor Antagonist, Bosentan on Patients With Poorly Controlled Asthma-A 17 Week, Double-blind, Placebo Controlled Crossover Trial
Brief Title: Bosentan for Poorly Controlled Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruitment.
Sponsor: UConn Health (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Mark Metersky, MD, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-287-1; 001
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Crossover (Other)
  Interventions: Drug: bosentan; Drug: placebo

INTERVENTIONS:
Drug: bosentan — Bosentan 62.5mg or placebo orally, twice a day for four weeks. After four weeks at this dose the subjects will have an increase to bosentan 125 mg or placebo orally twice daily for another four weeks. At week eight, subjects will crossover to bosentan or placebo depending upon their first randomization.
Drug: placebo — Bosentan 62.5mg or placebo orally, twice a day for four weeks. After four weeks at this dose the subjects will have an increase to bosentan 125 mg or placebo orally twice daily for another four weeks. At week eight, subjects will crossover to bosentan or placebo depending upon their first randomization.

SUMMARY:
Hypothesis: The endothelin-1 receptor antagonist, bosentan when added to the treatment of asthma patients who are symptomatic despite the use of controller therapy will improve asthma symptoms and physiology.

Twenty patients with a diagnosis of asthma, between the ages of 21 and 70 who are symptomatic despite the use of at least one controller medication will be randomized to either placebo or active medication for an 8 week period (initial 4 weeks is at 1/2 of final dose as per package insert and FDA approval). Measures of lung function and symptoms will be recorded. Patients will then cross over, so that patients initially on placebo will receive active drug for 8 weeks and those initially on active drug will receive placebo. The same endpoints will be measured. The acute bronchodilator effects of the drug will also be tested on the first day of therapy at the full therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, maintained on a minimum of 1 anti-inflammatory/controller and daily long acting B-agonist therapy with inadequate control of symptoms. (Defined as symptoms including wheezing, chest tightness or shortness of breath occurring at least 3 times a week or requiring use of "rescue" short-acting B-agonist at least 3 times a week).
* FEV1 less than 80% of predicted and greater than 40% at screening visit.
* A minimum of 12% reversibility of FEV1 after albuterol on screening visit or previously documented during the prior two years.
* Women of childbearing potential must use 2 non-hormonal methods of birth control (2 methods between the subject and her partner) while on the study and for 1 month after the last dose of study medication.
* Male subjects must use two non hormonal methods of birth control (2 methods between the subject and his partner) while on the study and for 1 month after the last dose of study medication.

Exclusion Criteria:

* History of liver disease, clinically significant cardiac disease, renal disease or pulmonary disease other than asthma. Patients with clinically significant laboratory abnormalities of LFTs/bilirubin (AST/ALT, TBili, alkaline phosphatase) and clinically significant anemia will be excluded. Clinically significant anemia will be defined as any anemia resulting in serum Hgb more than 1 gm/dl below the LLN, Patients with isolated minimal elevations of bilirubin (eg. as occurs in Gilbert's disease) or minimal elevations in transaminases (less than 1.2 x ULN) without a history of liver disease, risk factors for liver disease or symptoms of liver disease may still be included in the study at the investigator's discretion, but will have LFT testing at each study visit.)
* Cigarette history of >10 pack years.
* Predicted inability to adhere to medication regimen or documentation requirements of the study (symptom and medication diaries).
* Respiratory infection during 30 days preceding screening visit.
* Requirement for change in scheduled asthma medication use, including oral steroid dose change, or acute medical care for asthma during the 30 days preceding screening visit.
* Predicted inability to safely refrain from B-agonist use for the required amount of time on study visit days.
* Use of tiotropium
* Pregnancy, breast feeding or the use of hormonal methods of birth control as the only means of birth control during the study.
* Use of potent CYP3A4 and CYP2C9 inhibitors, including, but not limited to azole antifungals, amiodarone, glyburide, warfarin, cyclosporine, ritonavir, other medications potentially toxic to the liver or bone marrow.
* Use of any illegal drugs or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Metersky, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Bosentan 62.5mg or placebo orally, twice a day for four weeks. After four weeks at this dose the subjects will have an increase to bosentan 125 mg or placebo orally twice daily for another four weeks. At week eight, subjects will crossover to bosentan or placebo depending upon their first randomization.
Period: Overall Study
Arm/Group | All Study Participants
Started | 11
Completed | 7
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1
Time Frame: 1, 2, 4 hours after dosing
Measure: Mean (95% Confidence Interval); unit: liters
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 7 | 7
liters
  1 hour FEV1 | 1.50 [NA to NA] — Confidence interval not evaluable due to small number of participants | 1.57 [NA to NA] — Confidence interval not evaluable due to small number of participants
  2 hour FEV1 | 1.53 [NA to NA] — Confidence interval not evaluable due to small number of participants | 1.57 [NA to NA] — Confidence interval not evaluable due to small number of participants
  4 hour FEV1 | 1.50 [NA to NA] — Confidence interval not evaluable due to small number of participants | 1.51 [NA to NA] — Confidence interval not evaluable due to small number of participants

2. Primary Outcome: Peak Flow
Time Frame: last 7 days of each dosing period
Population: Data not analyzed, study terminated early
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Symptom Scores
Description: Symptom score could range from a minimum of 7 (no symptoms) to 35 (severe symptoms)
Time Frame: Last 7 days of each dosing period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 7 | 7
score on a scale | 19.7 (7.6) | 20.1 (3.5)

4. Secondary Outcome: FEV1
Time Frame: end of dosing period
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 7 | 7
liters | 1.46 (0.4) | 1.49 (0.47)

5. Secondary Outcome: Rescue Beta-agonist
Time Frame: end of each dosing period
Measure: Mean (Standard Deviation); unit: puffs of rescue inhaler
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 7 | 7
puffs of rescue inhaler | 34.6 (19.2) | 36.3 (18.9)

6. Other Pre Specified Outcome: Requirement for Escalation of Controller Medication.
Time Frame: 17 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Requirement for Urgent Medical Care for Asthma.
Time Frame: 17 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Ability to Taper Systemic Steroids Among Those Patients Who Are on Systemic Steroids at Study Entry.
Time Frame: 17 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Asthma Control Test Questionnaire
Description: Patient reported outcome minimum 5 (no symptoms) maximum 25 (severe symptoms)
Time Frame: end of each dosing period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Bosentan
Number analyzed (Participants) | 7 | 7
scores on a scale | 13.6 (5.0) | 13.1 (3.9)

ADVERSE EVENTS:
Time Frame: 17 weeks
Description: Non-Serious Adverse Events were not Analyzed, Terminated Study
Groups:
- Bosentan: Bosentan 62.5mg orally, twice a day for four weeks.
- Placebo: Placebo orally, twice a day for four weeks.
Arm/Group | Bosentan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/11
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan (N=9) | Placebo (N=11)
Abnormal liver function blood tests (Hepatobiliary disorders) | 0 (0) | 1 (1) — Very elevated liver function tests, while receiving placebo

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No